## **Evaluating ChatGPT-40, Gemini and Claude 3.7 in Endodontic Diagnostics:**

A Prospective Clinical Study

NCT number: not applicable

Ethical Approval: Date: 26.06.2025, Protocol No: 2025-07-02/38

Record Release Date/Time: November 24, 2025 14:03

Last Updated: December 8, 2025

## Statistical analysis

Data were entered into Excel and analyzed using SPSS (v27). Descriptive statistics were reported, and categorical comparisons were performed using Pearson chi-square or Fisher's Exact tests where appropriate, with a significance threshold of p < 0.05.